CLINICAL TRIAL: NCT05331027
Title: The Effect of Desflurane Versus Sevoflurane on Postoperative Recovery in Patients Undergoing Minor- to Moderate-risk Noncardiac Surgery - a Prospective Double-blinded Randomized Clinical Trial
Brief Title: The Effect of Desflurane Versus Sevoflurane on Postoperative Recovery
Acronym: RAPID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christian Reiterer, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RAPID_01
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Postoperative Recovery; Postoperative Delirium; Difference in Pharmakokinetics of Volatile Anesthetics
Keywords: Minor- to moderate-risk noncardiac surgery; Desflurane; Sevoflurane; Postoperative recovery
MeSH Terms: conditions — Emergence Delirium | interventions — Desflurane; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Desflurane Group (Experimental): After induction of anesthesia maintenance of anesthesia will be performed using goal-directed administration of desflurane with an intraoperative goal of bispectral index (BIS) 50±5.
  Interventions: Drug: Desflurane
- Sevoflurane Group (Active Comparator): After induction of anesthesia maintenance of anesthesia will be performed using goal-directed administration of sevoflurane with an intraoperative goal of bispectral index (BIS) 50±5.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Desflurane — After induction of anesthesia maintenance of anesthesia will be performed using goal-directed administration of desflurane with an intraoperative goal of bispectral index (BIS) 50±5.
  Arms: Desflurane Group
Drug: Sevoflurane — After induction of anesthesia maintenance of anesthesia will be performed using goal-directed administration of sevoflurane with an intraoperative goal of bispectral index (BIS) 50±5.
  Arms: Sevoflurane Group

SUMMARY:
Patients over the age of 65 years are at increased risk for developing delirium and cognitive complications in the immediate postoperative period after noncardiac surgeries, resulting in increased morbidity and mortality. Previous small studies have shown beneficial effects of desflurane on postoperative cognitive recovery, which has been explained by the more rapid onset and offset of anesthesia as compared to sevoflurane. However, there are very limited data on the effect of desflurane on postoperative recovery and time until criteria for discharge from post-anesthesia care unit (PACU) are fulfilled in elderly patients undergoing minor-to moderate-risk noncardiac surgery. Therefore, the investigators will test the primary hypothesis that general anesthesia with desflurane significantly reduces the time between discontinuation of volatile anesthetics after the end of surgery and reaching ready for discharge from PACU criteria, which are defined as reaching a modified Aldrete score ≥ 12, as compared to sevoflurane in patients ≥ 65 years of age undergoing minor-to moderate-risk noncardiac surgery.

DETAILED DESCRIPTION:
Background: Patients over the age of 65 years are at increased risk for developing delirium and cognitive complications in the immediate postoperative period after noncardiac surgeries, resulting in increased morbidity and mortality. Previous small studies have shown beneficial effects of desflurane on postoperative cognitive recovery, which has been explained by the more rapid onset and offset of anesthesia as compared to sevoflurane. However, there are very limited data on the effect of desflurane on postoperative recovery and time until criteria for discharge from post-anesthesia care unit (PACU) are fulfilled in elderly patients undergoing minor-to moderate-risk noncardiac surgery. Therefore, the investigators will test the primary hypothesis that general anesthesia with desflurane significantly reduces the time between discontinuation of volatile anesthetics after the end of surgery and reaching ready for discharge from PACU criteria, which are defined as reaching amodified Aldrete score ≥ 12, as compared to sevoflurane in patients ≥ 65 years of age undergoing minor-to moderate-risk noncardiac surgery.

Methods: The investigators will include 190 patients ≥ 65 years of age undergoing minor-to moderate-risk noncardiac surgery in this randomized, double-blinded clinical trial. Patients will be randomly assigned to receive desflurane or sevoflurane throughout surgery for maintenance of anesthesia. The primary outcome will be the time between discontinuation of desflurane until full postoperative recovery assessed via consecutive Aldrete Score assessments in the first 90 minutes after arrival at PACU. Aldrete Score will be assessed upon arrival at PACU and thereafter in five-minute intervals.

Statistics: The primary outcome, the time from discontinuation of volatile anesthetic agent to reaching discharge criteria from PACU assessed via Aldrete Score values,will be compared between both study groups using a Mann-Whitney-U test. Furthermore, the investigators will perform a median regression model for time to Aldrete score ≥ 12 points accounting for group as a factor as well as further covariables e.g. age, gender, weight.

Level of originality: Data regarding the effects of general anesthesia using desflurane in comparison to sevoflurane on postoperative recovery are mainly available from small studies. So far, there is very limited data on postoperative recovery and neurocognitive rehabilitation in elderly patients. However, this patient population is at a higher risk of developing postoperative neurocognitive complications, and could therefore, profit from a more rapid resurgence from anesthesia and postoperative recovery. Moreover, outpatient surgery will be becoming even more important. Therefore, reduction in postoperative PACU stay in combination with a decreased risk to develop postoperative delirium or cognitive dysfunction, might therefore improve outcome in this patient population as well.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 65 years of age at time of surgery
* Scheduled for elective minor- to moderate-risk noncardiac surgery with expected time of surgery ≤ 2 hours

Exclusion Criteria:

* Patients undergoing emergency surgery
* Patients undergoing bariatric surgery
* History of documented dementia / neurologic disorder
* Language, vision, or hearing impairments that may compromise cognitive assessments
* History of malignant hyperthermia
* History of structural muscle disease

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 190 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Modified Aldrete Score | Consecutive measurements until reaching 12 points for a maximum of 90 minutes after surgery and reaching PACU.
  A score to assess readiness of discharge from postanesthesia care unit (PACU). Patients can achieve 0-14 points in the modified Aldrete Score. A modified Aldrete Score > 12 points signals that criteria for discharge from PACU have been fulfilled, a modified Aldrete Score < 12 points signals that patients should stay in PACU.

SECONDARY OUTCOMES:
Secondary Outcome 1: Number of liters of supplemental oxygen administered in PACU for SpO2 ≥ 93% | Until reaching 12 points of the modified Aldrete score for a maximum of 90 minutes after surgery and reaching PACU.
  Postoperative need for administration of supplemental oxygen to maintain a SpO2 of ≥ 93% during PACU stay
Secondary Outcome 2: Postoperative cerebral oxygen saturation | Until reaching 12 points of the modified Aldrete score for a maximum of 90 minutes after surgery and reaching PACU.
  Postoperative non-invasive near-infrared spectroscopy for measurement of cerebral oxygenation
Secondary Outcome 3: Postoperative bispectral index values | Until reaching 12 points of the modified Aldrete score for a maximum of 90 minutes after surgery and reaching PACU.
  Postoperative continuous measurement of bispectral index for detection of postoperative aftereffects of anesthesia on awareness
Secondary Outcome 4: Ready for Hospital Discharge Scale Scores | For the first three postoperative days
  A score to evaluate patients' subjective readiness for hospital discharge. Patients can achieve 0-80 points in the Ready for Hospital Discharge Scale. Higher scores mean that patients are ready for hospital discharge, lower scores mean that patients are not ready for hospital discharge.

OTHER OUTCOMES:
Tertiary Outcome 1: NT-proBNP | Within the first two postoperative days
  Maximum concentrations of NT-proBNP
Tertiary Outcome 2: Troponin T | Within the first two postoperative days
  Maximum concentrations of Troponin T
Tertiary Outcome 3: Copeptin | Within the first two postoperative days
  Maximum concentrations of Copeptin
Tertiary Outcome 4: Interleukin-6 | Within the first two postoperative days
  Maximum concentrations of Interleukin-6
Tertiary Outcome 5: Procalcitonin | Within the first two postoperative days
  Maximum concentrations of Procalcitonin
Tertiary Outcome 6: CRP | Within the first two postoperative days
  Maximum concentrations of CRP
Tertiary Outcome 7: S100-B | Within the first two postoperative days
  Maximum concentration of S-100B
Exploratory Outcome 8: Delirium | For the first three postoperative days
  3D-CAM questionnaires for the evaluation of postoperative delirium. Patients can achieve 0-22 points in the 3D-CAM questionnaire. Higher scores indicate confusion, lower scores indicate no confusion.
Exploratory Outcome 9: Postoperative cognitive dysfunction | 30 days after surgery
  Montreal cognitive assessments for the evaluation of long-term postoperative cognitive dysfunction. Patients can achieve 0-22 points in the Montreal cognitive assessment. A reduction of 2 points from baseline indicates postoperative cognitive dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Reiterer, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
We will not share any individual participant data